CLINICAL TRIAL: NCT06958640
Title: Da Qing Offspring Study
Status: Enrolling by invitation | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Daqing Oil Field Hospital (Other)
Responsible Party: Principal Investigator, Bo Zhang, Professor, China-Japan Friendship Hospital
Other Study IDs: 2022-NHLHCRF-YS-01
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases (CVD); Offspring, Adult; Impaired Glucose Tolerance (Prediabetes); Prevention; Cancer; Comorbidity; Inter- and Transgenerational Inheritance
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Glucose Intolerance; Prediabetic State; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lifestyle intervention subjects and offspring group: The subjects who received lifestyle intervention in the original Daqing Diabetes Prevention Study, their spouses, children 1 to 3, and spouses of their offspring were included in the study.
  Interventions: Behavioral: Lifestyle interventions
- Control group subjects and offspring: The subjects who did not received lifestyle intervention in the original Daqing Diabetes Prevention Study, their spouses, children 1 to 3, and spouses of their offspring were included in the study.

INTERVENTIONS:
Behavioral: Lifestyle interventions — Dietary intervention: 30kcal energy intake per kilogram of body weight per day, increase vegetable intake, control sugar and alcohol intake, encourage overweight and obese people to lose weight, lose 0.5-1kg per month until the weight reaches the target.
  Exercise intervention: Appropriate physical activity in spare time, 30-40 minutes per day, 5 times a week.
  Groups: Lifestyle intervention subjects and offspring group

SUMMARY:
This is an observational study tracking families and offspring of three cohorts from the 1986 Da Qing study: newly diagnosed diabetes, impaired glucose tolerance, and normoglycemia groups. Based on the original participants, the study will further include their spouses, first to third-generation offspring, and spouses of the offspring. General demographic information will be collected, and anthropometric measurements will be refined. A structured questionnaire will be used to gather disease history, family history of diabetes, and related information. Comprehensive diabetes-related laboratory screening and complication assessments will be conducted. A standardized biobank will be established, including blood and urine samples from the Da Qing Offspring Study, to support future research on epigenetics, metabolomics, and other mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Spouses of the original Daqing diabetes Prevention Research Population (IGT), offspring 1 to 3 generations, and offspring spouses were included in the study, without special restrictions on subjects' gender, age, basic disease status, etc。
* Conduct a death agent investigation for some deceased members.

Exclusion Criteria:

▪People who are unwilling to participate in this study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Original subjects and spouses (70-90 years old), N=576+576=1152; First generation (50-70 years old), based on an average of 3 children per family, N=576*3=1728; The marriage rate of first generation is 90%, and the spouses N=1555; Second generation (25-45 years old), based on 90% of families having children, with an average of 1 child per family, N=1555*90%*1=1400; The marriage rate of second generation is 70%, and the spouses N=1400*70%=980; Third generation (1-20 years old), based on 80% of families having children, with an average of 1 child per family, N=980*80%*1=784; Based on the follow-up rate of 70%, the total number of people is about 5,000.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of diabetes | Through study completion, an average of about 1.5 years
  This study statistically analyzed the cumulative incidence rate of diabetes at the end of the study through interview, medical record review, physical examination

SECONDARY OUTCOMES:
weight | Through study completion, an average of about 1.5 years
  The subject's weight is recorded and the results are reported in kilograms.
waist circumference | Through study completion, an average of about 1.5 years
  The subjects' waist circumference was recorded and the waist circumference results were reported in centimeters.
Height | Through study completion, an average of about 1.5 years
  The subject's height was recorded, and the results were recorded in centimeters.
Exercise frequency and intensity | Through study completion, an average of about 1.5 years
  The subjects' daily exercise frequency and intensity were recorded.
Coronary heart disease incidence | Through study completion, an average of about 1.5 years
  This study statistically analyzed the incidence of coronary heart disease at the end of the study through interview, medical record review, physical examination
all-cause deaths | Through study completion, an average of about 1.5 years
  This study counted all-cause deaths at the end of the study through death certificate, medical record review, family interview
incidence of diabetic peripheral neuropathy | Through study completion, an average of about 1.5 years
  This study statistically analyzed the incidence of diabetic peripheral neuropathy at the end of the study through interview, medical record review, physical examination
other cause mortality | Through study completion, an average of about 1.5 years
  This study statistically analyzed other cause mortality at the end of the study through death record, medical record review, family interview
cardiovascular mortality rate | Through study completion, an average of about 1.5 years
  This study statistically analyzed the cardiovascular mortality rate at the end of the study through death certificate, medical record review, family interview
incidence of blindness | Through study completion, an average of about 1.5 years
  This study statistically analyzed the incidence of blindness at the end of the study through interview, medical record review, physical examination
Diabetic retinopathy incidence | Through study completion, an average of about 1.5 years
  This study statistically analyzed the incidence of diabetic retinopathy at the end of the study through interview, medical record review, physical examination
Diabetic nephropathy incidence | Through study completion, an average of about 1.5 years
  This study statistically analyzed the incidence of diabetic nephropathy at the end of the study through interview, medical record review, physical examination
Peripheral vascular disease incidence | Through study completion, an average of about 1.5 years
  This study statistically analyzed the incidence of peripheral vascular disease at the end of the study through interview, medical record review, physical examination
Heart failure incidence | Through study completion, an average of about 1.5 years
  This study statistically analyzed the incidence of heart failure at the end of the study through interview, medical record review, physical examination
Stroke incidence | Through study completion, an average of about 1.5 years
  This study statistically analyzed the incidence of stroke at the end of the study through interview, medical record review, physical examination
dietary habits | Through study completion, an average of about 1.5 years
  The subjects' eating habits and dietary preferences were assessed through patient interviews.
health-related quality of life | Through study completion, an average of about 1.5 years
  The EuroQol questionnaire or health status questionnaire was administered through patient interviews to assess the subjects' health-related quality of life.
blood pressure | Through study completion, an average of about 1.5 years
  During the visit, the subjects' systolic and diastolic blood pressures were measured at rest by physical examination. The measurements were performed twice and the average was taken.
blood sugar | Through study completion, an average of about 1.5 years
  Blood samples were collected from the subjects at 1 hour and 2 hours after the steamed bread meal when they were fasting. The blood samples were used to test blood sugar levels and blood lipids, including total cholesterol, triglycerides, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol.
blood lipid | Through study completion, an average of about 1.5 years
  Venous blood was collected from the subjects in a fasting state. The blood samples were used to test blood lipid status, including total cholesterol, triglycerides, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol.
skin AGE | Through study completion, an average of about 1.5 years
  The skin AGE of the subjects was measured by physical examination. After cleaning the inner skin of the forearm, the AGE Reader probe was gently placed on the skin surface, the excitation light was emitted and the fluorescence intensity was recorded. The results were repeated 3 times and the average value was taken.
Tidal Volume | Through study completion, an average of about 1.5 years
  The subjects were assessed for Tidal Volume, which reflects the ventilation efficiency in the basic breathing state. Tidal Volume is measured in liters.
Functional Residual Capacity | Through study completion, an average of about 1.5 years
  Subjects were assessed for Functional Residual Capacity, which reflects lung capacity. Functional Residual Capacity is measured in liters.
Forced Vital Capacity | Through study completion, an average of about 1.5 years
  The subjects were assessed for Forced Vital Capacity, which reflects the overall ventilation capacity of the lungs. Forced Vital Capacity is measured in liters.
Forced Expiratory Volume in 1 second | Through study completion, an average of about 1.5 years
  The subjects were assessed for Forced Expiratory Volume in 1 second, which reflects respiratory reserve capacity. Forced Expiratory Volume in 1 second is measured in liters.

CONTACTS AND LOCATIONS:
Overall Officials: Liping Yu, Doctor, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lindstrom J, Ilanne-Parikka P, Peltonen M, Aunola S, Eriksson JG, Hemio K, Hamalainen H, Harkonen P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Mannelin M, Paturi M, Sundvall J, Valle TT, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Sustained reduction in the incidence of type 2 diabetes by lifestyle intervention: follow-up of the Finnish Diabetes Prevention Study. Lancet. 2006 Nov 11;368(9548):1673-9. doi: 10.1016/S0140-6736(06)69701-8. PMID 17098085
- [Background] Sakane N, Sato J, Tsushita K, Tsujii S, Kotani K, Tsuzaki K, Tominaga M, Kawazu S, Sato Y, Usui T, Kamae I, Yoshida T, Kiyohara Y, Sato S, Kuzuya H; Japan Diabetes Prevention Program (JDPP) Research Group. Prevention of type 2 diabetes in a primary healthcare setting: three-year results of lifestyle intervention in Japanese subjects with impaired glucose tolerance. BMC Public Health. 2011 Jan 17;11(1):40. doi: 10.1186/1471-2458-11-40. PMID 21235825
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Gong Q, Zhang P, Wang J, Ma J, An Y, Chen Y, Zhang B, Feng X, Li H, Chen X, Cheng YJ, Gregg EW, Hu Y, Bennett PH, Li G; Da Qing Diabetes Prevention Study Group. Morbidity and mortality after lifestyle intervention for people with impaired glucose tolerance: 30-year results of the Da Qing Diabetes Prevention Outcome Study. Lancet Diabetes Endocrinol. 2019 Jun;7(6):452-461. doi: 10.1016/S2213-8587(19)30093-2. Epub 2019 Apr 26. PMID 31036503
- [Background] Gong Q, Zhang P, Wang J, Gregg EW, Cheng YJ, Li G, Bennett PH; Da Qing Diabetes Prevention Outcome Study Group. Efficacy of lifestyle intervention in adults with impaired glucose tolerance with and without impaired fasting plasma glucose: A post hoc analysis of Da Qing Diabetes Prevention Outcome Study. Diabetes Obes Metab. 2021 Oct;23(10):2385-2394. doi: 10.1111/dom.14481. Epub 2021 Jul 27. PMID 34212465